CLINICAL TRIAL: NCT06101615
Title: Effects of Instrument Assisted Soft Tissue Mobilization vs. Foam Rolling on Knee and Hip Flexibility and Performance in Soccer Players
Brief Title: Effects of IASTM vs. Foam Rolling on Knee and Hip Range of Motion in Soccer Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01616 Mansoor Kh Achakzai
Record Dates: First submitted 2023-10-11; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Muscle Tightness
Keywords: FAT; Foam Rolling; IASTM; Joint Flexibility; Soccer

STUDY DESIGN:
Intervention Model Description: Concurrent Parallel Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): IASTM Group
  Interventions: Other: IASTM (FAT)
- Group B (Active Comparator): Foam Rolling Group
  Interventions: Other: Foam Rolling

INTERVENTIONS:
Other: IASTM (FAT) — Group-A participants would receive Facial Abrasion Technique (FAT) with an Instrument, FAT-Tool. Treatment sessions will be carried out three times per week for eight weeks after an initial warm-up session. All the sessions will be performed at the same time of day (i.e., between 4-6 pm), to avoid possible confounding circadian effects. The FAT group will receive 2 min application on the quadriceps and hamstring muscles with a FAT-tool Pro Large model, which consists of a handle and 20cm treatment surface. The muscles will be treated in a pre-stretched position, meaning a knee flexion in a supine position for the quadriceps muscle and a hip flexion and knee extension in a side-lying position for the hamstring muscles.
  Arms: Group A
Other: Foam Rolling — Group-B participants would receive Foam Rolling (FR). Treatment sessions will be carried out three times per week for eight weeks after an initial warm-up session. All the sessions will be performed at the same time of day (i.e., between 4-6 pm) to avoid possible confounding circadian effects. The Foam Roller group will receive 2x1 min of FR on the quadriceps and the hamstrings on the dominant leg with the opposite leg crossed over the dominant one. During each minute the muscle will be rolled out 4-5 times, with a break of 30s in between sets. They will be instructed to utilize short, kneading like movements in one direction and a quick motion in the other direction. A grid foam roller will be utilized with a length of 33cm, diameter of 14 cm and with a hard hollow core, wrapped in ethylene vinyl acetate foam.
  Arms: Group B

SUMMARY:
The aim of this study is:

To compare the acute and long-term affects of instrument assisted soft tissue mobilization (IASTM) vs foam rolling on knee and hip flexibility and performance in soccer players.

DETAILED DESCRIPTION:
The objective of this study is to compare the acute and long-term affects of instrument assisted soft tissue mobilization vs foam rolling on knee and hip flexibility and performance in soccer players. This is a randomized controlled trial, in which participants will be randomly divided into two groups: group-A and group-B. Group-A will receive intervention IASTM while Group-B will receive foam rolling as intervention. Intervention will be carried out for 8 weeks. Assessment of the range of motions for hip and knee joints will be carried out at baseline, immediately after the session, after four weeks and after five (5) months. The secondary measures of performance used in the study are sit and reach test, 100m sprint speed test, Illinois agility run test.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with normal BMI
* Players with at least one year of playing professional soccer and taking at least three training sessions/matches per week.

Exclusion Criteria:

* Players with any pathological conditions affecting any of the system.
* Suffering from recent acute unhealed MSK injury/Trauma.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Knee Range of Motion (ROM) | Baseline, after 8 weeks, and after 5 months
  Knee ROM will be measured using universal goniometer.

SECONDARY OUTCOMES:
Knee Flexibility (Active Knee Extension Test) | Baseline, after 8 weeks, and after 5 months
  Knee flexibility will be assessed using the Active Knee Extension (AKE) test. Assessment of this test will be carried out through a universal goniometer.
Knee Flexibility (Sit and Reach Test) | Baseline, after 8 weeks, and after 5 months
  Knee flexibility will also be assessed using the Sit and Reach Test. Assessment of this test will be carried out through an improvised ruler/measuring tape.
Sprint Speed | Baseline, after 8 weeks, and after 5 months
  Sprint speed will be assessed using the time required to complete 100m Sprint Test.
Agility | Baseline, after 8 weeks, and after 5 months
  Agility will be measured using the time required to complete the Illinois Agility Run Test (IART).

CONTACTS AND LOCATIONS:
Overall Officials: Noman Sadiq, MS-SPT, Principal Investigator — Riphah International University, Islamabad.
Locations (1):
- Riphah International University (RIU), Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No